CLINICAL TRIAL: NCT06658652
Title: A Clinical Study to Evaluate the Effect of Food and Water Volume on the Pharmacokinetics of the MK-0616 Final Market Formulation in Healthy Adult Participants
Brief Title: The Effect of Food and Water Volume in Healthy Adult Participants Administered Enlicitide Decanoate (MK-0616) (MK-0616-022)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0616-022; MK-0616 (Other: MSD)
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — MK-0616

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Enlicitide Decanoate Food Effect (Experimental): Participants will be administered enlicitide decanoate on Day 1 with or without food.
  Interventions: Drug: Enlicitide decanoate
- Enlicitide Decanoate Water Effect (Experimental): Participants will be administered enlicitide decanoate on Day 1 with high, medium, and low volumes of water.
  Interventions: Drug: Enlicitide decanoate

INTERVENTIONS:
Drug: Enlicitide decanoate — Oral tablet
  Other Names: MK-0616

SUMMARY:
Enlicitide decanoate (MK-0616, the study medicine) is in a class of medicines that have been shown to reduce LDL-C. Enlicitide decanoate is different from the other medicines in this class because it is taken as a tablet and not an injection.

The goal of this study is to see what happens to doses of enlicitide decanoate in a person's body over time. During the study, researchers will measure people's blood samples for the amount of enlicitide decanoate when taken with food or on an empty stomach, or when taken with high, medium, and low volumes of water. Researchers also want to learn about the safety of enlicitide decanoate, including how well people tolerate (manage) it.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2
* Is medically healthy with no clinically significant medical history

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has history of gastrointestinal disease which may affect food and drug absorption
* Has history of cancer (malignancy).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-24 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the AUC0-Inf of enlicitide decanoate.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of Enlicitide Decanoate | Pre-dose and at designated time points up to 24 hours postdose
  Blood samples will be collected to determine the AUC0-24 of enlicitide decanoate.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the AUC0-last of enlicitide decanoate.
Maximum Plasma Concentration (Cmax) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the Cmax of enlicitide decanoate.
Time to Maximum Plasma Concentration (Tmax) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the Tmax of enlicitide decanoate.
Lag Time (tlag) of Enlicitide Decanoate in Plasma | Pre-dose and at designated time points up to 1 week postdose
  Tlag is the time from dosing to the first appearance in plasma. Blood samples will be collected to determine the tlag of enlicitide decanoate.
Apparent Terminal Half-life (t1/2) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the t1/2 of enlicitide decanoate.
Apparent Clearance (CL/F) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the CL/F of enlicitide decanoate.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Enlicitide Decanoate | Pre-dose and at designated time points up to 1 week postdose
  Blood samples will be collected to determine the Vz/F of enlicitide decanoate.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to 14 days postdose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to 14 days postdose
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com